CLINICAL TRIAL: NCT04316533
Title: Study of the Association Between Work Stress and the Impact of Pruritus on Quality of Life
Brief Title: Work Stress and Impact of Pruritus on Quality of Life
Acronym: PRUERI
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC19.0263
Record Dates: First submitted 2020-03-06; First posted 2020-03-20 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Psoriasis
Keywords: Psoriasis; Occupational stress; Pruritus; Quality of life
MeSH Terms: conditions — Psoriasis; Occupational Stress; Pruritus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Work stress and pruritus: imbalance of effort balance reward in patients with psoriasis.

DETAILED DESCRIPTION:
Background. Stress increases the likelihood of psoriasis flare-up episodes and itching. Few studies have focused on work-related stress on such skin symptoms.

Objective. To study the association between work-related stress, pruritus and quality of life among workers suffering from psoriasis.

Methods. Investigators will conduct a monocentric non-interventional prospective study. Patients suffering from psoriasis will be recruited in both the Dermatology inpatient ward and outpatient clinic of Brest University Hospital . Included patients will be workers. Work-related stress will be assessed using the Effort-Reward Imbalance (ERI) model. The impact of pruritus on quality of life will be assessed with the Itchy Quality of Life (ItchyQoL) self-administered questionnaire. The collected data will include age, sex, body mass index, ordered medication to treat psoriasis, weekly working hours. The association between ERI and ItchyQoL scores will be studied using a univariate logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* Major patients
* Active busy patients with psoriasis presenting for a dermatology consultation or hospitalization at the Brest CHRU
* Participation agreement

Exclusion Criteria:

* Presence of another potentially pruritic pathology
* No command of the French language
* Patient under legal protection (guardianship, curatorship, etc.)
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Active and employed population, suffering from psoriasis, presenting for consultation or hospitalization of dermatology at the CHRU of Brest
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Pruritus' impact on quality of life | time required to complete the self questionnaire estimated at approximately 5 min immediately after consultation with the dermatologist
  The Itchy Quality of Life questionnaire (ItchyQoL) assess the quality of life linked to pruritus. It is a 22-item questionnaire wich assess the frequency of pruritus'symptoms in the past seven days. The score is between 22 and 110. The higher the score, the greater the impact of pruritus.

SECONDARY OUTCOMES:
Occupational stress | time required to complete the self questionnaire estimated at approximately 5 min immediately after consultation with the dermatologist
  The effort-reward imbalance questionnaire in 23-item for occupational stress. Six items make it possible to calculate the extrinsic efforts felt (score e) and eleven items assess the rewards perceived by the employee (score r). The ERI score is then calculated as follows: Ratio = (11 x e) / (6 x (66 - r)) (e: effort scale score, r: rewards scale score). A ratio greater than one indicates an imbalance in favor of efforts. The last six items make it possible to calculate the score for intrinsic efforts (over commitement). They relate to the inability to get away from work, impatience and disproportionate irritability.

CONTACTS AND LOCATIONS:
Locations (1):
- Chru Brest, Brest, Finistère, France